CLINICAL TRIAL: NCT02915237
Title: Development of a Polyphenol-rich Dietary Preparation for Treating Veterans With Gulf War Illness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Department of Veterans Affairs, New Jersey (U.S. Federal Agency)
Responsible Party: Principal Investigator, Giulio Maria Pasinetti, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 13-1398
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Gulf War Illness
Keywords: Veterans; Gulf War Illness; Gulf War Veterans's Illness; Gulf War Veterans' Medically Unexplained Illnesses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low Dose - Concord grape juice (Experimental): Daily dietary supplementation with 4 oz. of a commercially available Concord grape juice.
  Interventions: Dietary Supplement: Concord grape juice
- Moderate Dose - Concord grape juice (Experimental): Daily dietary supplementation with 8 oz. of a commercially available Concord grape juice.
  Interventions: Dietary Supplement: Concord grape juice
- High Dose - Concord grape juice (Experimental): Daily dietary supplementation with 16 oz. of a commercially available Concord grape juice.
  Interventions: Dietary Supplement: Concord grape juice
- Low dose - placebo beverage (Placebo Comparator): Daily dietary supplementation with 4 oz. of a placebo beverage
  Interventions: Dietary Supplement: Placebo Beverage
- Moderate Dose - placebo beverage (Placebo Comparator): Daily dietary supplementation with 8 oz. of a placebo beverage
  Interventions: Dietary Supplement: Placebo Beverage
- High Dose - placebo beverage (Placebo Comparator): Daily dietary supplementation with 16 oz. of a placebo beverage
  Interventions: Dietary Supplement: Placebo Beverage

INTERVENTIONS:
Dietary Supplement: Concord grape juice — Daily dietary supplementation with a commercially available Concord grape juice.
  Arms: High Dose - Concord grape juice; Low Dose - Concord grape juice; Moderate Dose - Concord grape juice
Dietary Supplement: Placebo Beverage — Daily dietary supplementation with a placebo beverage consisting of water, sugar, artificial flavoring and color that is formulated to look and taste like grape juice and have the same carbohydrate composition and energy load.
  Arms: High Dose - placebo beverage; Low dose - placebo beverage; Moderate Dose - placebo beverage

SUMMARY:
Gulf War Illness (GWI) is a multi-symptom disorder that is characterized by complex traits such as fatigue, headaches, joint pain, insomnia, and memory problems. With no treatment for GWI currently available, there is an urgent need to develop novel interventions to alleviate major GWI clinical complications. Recent evidence highlights the potential value of flavonoids, a subclass of organic chemical called polyphenols abundantly found in some plants and common dietary preparations, in helping relieve clinical complications in Veterans with GWI. The overall goal is to test whether daily consumption of commercially available Concord grape juice, which is very Flavonoid-rich, is effective for treating cognitive deficits and chronic fatigue in Veterans with GWI.

DETAILED DESCRIPTION:
Gulf War Illness (GWI) is a multi-symptom disorder that is characterized by complex traits. Clinical complications of GWI typically persist over long-term, cause significant pain and suffering, and interfere with the ability of affected Veterans to successfully integrate back into civilian society. There is no treatment for GWI and there is an urgent need to develop novel interventions either to resolve underlying GWI mechanisms, or to alleviate major GWI clinical complications.

Recent Evidence highlights the potential value of flavonoids, a subclass of organic chemical called polyphenols that are abundantly found in some plants and common dietary preparations may help alleviate chronic fatigue and preserve cognitive functions. Based on this, the overall goal is to test whether the potential efficacy of dietary supplementation with a commercially available flavonoid-rich product, alleviates clinical complications in Veterans with GWI. In particular, the researchers propose a randomized, double-blind, placebo-controlled Phase I/IIA study to test the feasibility and potential efficacy of Concord grape juice dietary supplementation to treat cognitive deficits and chronic fatigue in Veterans with GWI.

ELIGIBILITY:
Inclusion Criteria:

* Gulf War Veterans deployed to the Persian Gulf theatre between August 1990 and August 1991. GWI will be defined according to the Kansas Case Definition. The Kansas Case Definition identifies 6 symptom domains and requires endorsement of moderately severe and/or multiple symptoms in at least 3 of those domains. To meet the case definition, the Veterans must also indicate that each symptom first became problematic during or within one year of the Gulf War.

Exclusion Criteria:

* Individuals not meeting the inclusion criteria for Gulf War deployment and definition of GWI, or with conditions that might interfere with their ability to report their symptoms (e.g., drug use) are excluded.
* Additional exclusion criteria are current medical conditions that may explain the symptoms (diabetes, heart disease, among others) or significant current (in the past six months) unstable (requiring significant medication adjustments or hospitalization) psychiatric conditions, including suicidal or homicidal ideation, schizophrenia or bipolar disorder according to subject responses to the interview and review by the principal investigator.
* Subjects who usually consume abnormally high contents of dietary polyphenol based on a self-reported diet diary will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08; Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Brief Symptom Inventory (BSI) | 6 months
  to assess safety and tolerability to treatment. The test is a 53-item self report scale that uses the 5 point Likert scale.
Patient Health Questionnaire-15 (PHQ-15) | 6 months
  to assess safety and tolerability to treatment. The Patient Health Questionnaire 15 (PHQ 15) is a validated measure of somatic symptom severity in functional somatic syndromes (FSS). Scale ranges from 0-30 (mild to severe).
California Verbal Learning Test-Second Edition (CVLT-II) | 6 months
  This test looks at cognitive functioning by assessing immediate recall and long-delayed recall.
The Chalder Fatigue Questionnaire | 6 months
  The Chalder Fatigue Questionnaire assess chronic fatigue. Each of the 11 items are answered on a 4-point scale ranging from the asymptomatic to maximum symptomology

SECONDARY OUTCOMES:
Wechsler Adult Intelligence Scale (WAIS-IV) | 6 months
  The Digit Span subtest is a widely used measure of auditory attention that is well-normed and sensitive. The subtest has three parts - digits forward, backward, and sequencing.
the Conner's Continuous Performance Test-3 (CPT-3) | 6 months
  The CPT-3 assist in clinical assessment of attention problems. The patient is instructed to press the space bar (or mouse button) immediately following the presentation of specific letters on screen. The test normally takes 14 minutes to administer.
the Trail Making Test (TMT) | 6 months
  The TMT consists of two forms, parts A and B. This measure taps both simple graphomotor speed (Part A) and adds in a rapid set-shifting paradigm that taps executive functioning (Part B).
Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) Block Design Subtest | 6 months
  A tool for testing adult intelligence level.
the Stroop Test | 6 months
  The Stroop Color and Word Test consists of a Word Page with color words printed in black ink, a Color Page with 'Xs' printed in color, and a color-Word Page with words from the first page printed in colors from the second page (the color and the word do not match). The respondent goes down each sheet reading words or naming the ink colors as quickly as possible within a time limit. The test yields three scores based on the number of items completed on each of the three stimulus sheets. An Interference score, which is useful in determining the individual's cognitive flexibility, creativity, and reaction to cognitive pressures also can be calculated.
Halstead Category Test | 6 months
  This test takes approximately 30 minutes and consists of 120 items, presented visually. The participant must decipher the underlying principle of the stimulus set. Total number of errors will be used.
Brief Visuospatial Memory Test-Revised (BVMT-R) | 6 months
  A tool to measure visuospatial learning and memory abilities.
Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) Digit Span Subtest | 6 months
  Digit Span measures short-term auditory memory and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maria Pasinetti, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Brett Chaney, MD, Study Director — United States Department of Defense
Locations (1):
- VA- New Jersey Health Care System, East Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steele L. Prevalence and patterns of Gulf War illness in Kansas veterans: association of symptoms with characteristics of person, place, and time of military service. Am J Epidemiol. 2000 Nov 15;152(10):992-1002. doi: 10.1093/aje/152.10.992. PMID 11092441
- [Background] Helmer DA, Van Doren WW, Litke DR, Tseng CL, Ho L, Osinubi O, Pasinetti GM. Safety, Tolerability and Efficacy of Dietary Supplementation with Concord Grape Juice in Gulf War Veterans with Gulf War Illness: A Phase I/IIA, Randomized, Double-Blind, Placebo-Controlled Trial. Int J Environ Res Public Health. 2020 May 19;17(10):3546. doi: 10.3390/ijerph17103546. PMID 32438639
- See also: Web link for research studies that are open to Gulf War Veteran research at the New Jersey War Related Illness and Injury Study Center — https://urldefense.proofpoint.com/v2/url?u=http-3A__www.warrelatedillness.va.gov_WARRELATEDILLNESS_research_volunteer_nj-2Dwriisc.asp&d=AwIGaQ&c=4R1YgkJNMyVWjMjneTwN5tJRn8m8VqTSNCjYLg1wNX4&r=j-Ik801LfpKr-w6-cs0wCg&m=Axgk1UrBTBGADl2K9uFvA9a5vk96rKXyS_g718Wb_Yk&s=205Ow4GZ9bw3_awAAlmqGFf7BUAdXN2h9Jbi02KQmDw&e=